CLINICAL TRIAL: NCT06382402
Title: Randomized Control Trial of Outcomes Comparing a Coronary Computed Tomography Angiography (CCTA) Guided Management Strategy Versus a Standard of Care Strategy in Type 2 Non-ST-elevation MI
Brief Title: A CCTA Guided Management Strategy Versus a Standard of Care Strategy in Type 2 NSTEMI
Status: Withdrawn | Type: Observational
Why Stopped: study withdrawn, no participant enrolled, change in the study design planned
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Dinesh Kalra, MD, Professor, University of Louisville
Other Study IDs: 23.0924
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CCTA Group: CT group will undergo CCTA to evaluate for coronary artery disease to early address underlying CAD and then care will be directed based on the findings of that CT scan.
  Interventions: Radiation: CCTA scan
- No CCTA Group: Group 2 will not undergo CCTA and will be managed at the discretion of the primary team using the standard of care pathway comprising of either conservative medical management, stress testing, or invasive evaluation with coronary angiography in the catheterization laboratory.

INTERVENTIONS:
Radiation: CCTA scan — • CCTA will be performed per the standard clinical protocol using a Cannon Aquilion ONE scanner with 16 cm z-axis coverage at 0.5 mm resolution, low contrast, and reduced radiation dose requirements.
  Groups: CCTA Group

SUMMARY:
This study design is a prospective randomized control trial to compare outcomes between the utilization of coronary computed tomography angiography (CCTA) vs conservative treatment in type 2 NSTEMI. The targeted population is expectedly heterogeneous and inpatient setting who are admitted and diagnosed with type 2 NSTEMI.

DETAILED DESCRIPTION:
This study design is a prospective randomized control trial to compare outcomes between the utilization of coronary computed tomography angiography (CCTA) vs conservative treatment in type 2 NSTEMI. The targeted population is expectedly heterogeneous and inpatient setting who are admitted and diagnosed with type 2 NSTEMI. Patients are randomized into 2 groups. Group 1 undergoes coronary 64-detector row computed tomography angiography (CCTA) and Group 2 receives conservative management and treatment for underlying conditions. The investigators will evaluate cross-sectional and time-varying clinical, laboratory, and imaging characteristics in association with clinical events. The exclusion criteria are an absence of information for follow-up of clinical events, and patients who have absolute and relative contraindications for CCTA. Absolute contraindications are a patient history of severe or anaphylactic reaction to iodinated contrast, inability to cooperate with scan protocols, hemodynamic instability, decompensated heart failure, acute myocardial infarction, and renal impairment with GFR < 30. Relative contraindications include pregnancy, inability to tolerate heart rate-slowing medications or nitroglycerin, recent phosphodiesterase inhibitor use, severe aortic stenosis, bronchospastic disease, and patient's weight and height.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with type 2 NSTEMI
* Aged 18-70 years old
* At the University of Louisville and Jewish hospitals

Exclusion Criteria:

* History of severe or anaphylactic reaction to iodinated contrast
* Inability to cooperate with scan protocols
* Hemodynamic instability
* Decompensated heart failure
* Acute myocardial infarction
* Renal impairment with GFR < 30
* Pregnancy
* Inability to tolerate heart rate-slowing medications or nitroglycerin
* Recent phosphodiesterase inhibitor use
* Severe aortic stenosis
* Bronchospastic disease
* Patient's weight and height

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients diagnosed with type 2 NSTEMI.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
MACE | anytime within 3 years
  Time to the first major adverse cardiac event (MACE) at 3 years between 2 groups.
  Unit: no unit (yes/no)
Cardiovascular (CV) mortality | anytime within 3 years
  Cardiovascular (CV) mortality Unit: no unit (yes/no)
Nonfatal MI, stroke | anytime within 3 years
  Nonfatal MI, stroke Unit: no unit (yes or no)
Hospitalization for unstable angina | anytime within 3 years
  Hospitalization for unstable angina Unit: no unit (yes or no)
Hospitalization for heart failure | anytime within 3 years
  Hospitalization for heart failure Unit: no unit (yes or no)
Unplanned revascularization | anytime within 3 years
  Unplanned revascularization Unit: no unit (yes or no)

SECONDARY OUTCOMES:
All-cause mortality | anytime within 3 years
  All-cause mortality Unit: no unit (yes or no)
In-hospital and 90-day costs | anytime within 90 days
  In-hospital and 90-day costs Unit: US dollars
Patient quality of life at 90 days | anytime within 90 days
  Patient quality of life at 90 days Unit: The numeric rating scales
Diagnostic certainty scores | anytime within 3 years
  Diagnostic certainty scores Unit: The numeric rating scores
Individual components of the primary endpoint | anytime within 3 years
  Individual components of the primary endpoint Unit: no unit (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kalra, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville School of Medicine, Division of Cardiovascular Diseases, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No